CLINICAL TRIAL: NCT03975725
Title: Evaluation of an Ultraportable ECG Recording Device and Its Visualization Software for the Detection of Atrial Fibrillation
Acronym: WITCARD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-67; 2019-A00918-49 (Other: idrcb)
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Cardiovascular Illnesses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- witcard (Experimental)
  Interventions: Device: the use of the WitCard; Other: the use of WitDisplayer

INTERVENTIONS:
Device: the use of the WitCard — electrocardiogram (ECG)
Other: the use of WitDisplayer — a software to visualize, measure, annotate, comment, archive, and share the different ECGs acquired with the WitCard (ECGW) of different patients.

SUMMARY:
The purpose is to demonstrate the usefulness of WitCard and WitDisplayer in the diagnosis of AF but more generally in the qualification of the heart rhythm and the diagnosis of cardiac arrhythmias.

The main objective is therefore to demonstrate that at least 90 +/- 0.03% of ECGWs are interpretable by a physician and the primary endpoint will therefore be the ratio of the number of ECGWs that allowed a physician to make a diagnosis. rhythmic (ECGW interpretable) and the total number of ECGW recorded and viewed.

The clinical trial as part of the CE medical device certification process for secondary objectives and ancillary studies will be required to assess the diagnostic performance of the WitCard + WitDisplayer system, the quality of the ECGW recorded by the WitCard, the the safety of using the WitCard, the technical performance of the WitCard ECG recorder, the ergonomics of the WitCard, and finally the performance of automatic cardiac rhythm classification algorithms.

DETAILED DESCRIPTION:
Monocentric, prospective, interventional study

ELIGIBILITY:
Inclusion Criteria:

Patient, male or female, over 18 years of age, presenting to the cardiology-rhythmology department (consultations and hospitalizations) or to the emergency department of the Timone 2 Hospital for the management of suspicion of disorder heart rate in front of:

* Palpitations
* Dyspnoea, acute pulmonary edema, non-ischemic heart failure
* Malaise, lipothymia, syncope

Exclusion Criteria:

* Patients with clinical criteria that do not warrant the use of WitCard:
* Immediate vital risk whatever its nature
* Rhythmic urgency requiring treatment without delay: respiratory, circulatory or neurological distress
* Acute Coronary Syndrome
* Pregnant women
* Non-beneficiaries of a social security scheme
* Persons deprived of their liberty
* Patient participating in another study
* Patient in a period of exclusion determined by a previous study
* Patient under the protection of justice, under guardianship or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
the ratio between the number of ECGWs that allowed a physician to make a rhythmic diagnosis (ECGW interpretable) and the total number of ECGWs recorded and visualized. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille